CLINICAL TRIAL: NCT01456429
Title: Assessment of Surgical Mediastinal sTaging Added to Endoscopic Ultrasound in cN1 Lung canceR.
Brief Title: Assessment of Invasive Mediastinal Staging in cN1 Lung Cancer.
Acronym: ASTER2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Aster2-2010
Record Dates: First submitted 2011-10-18; First posted 2011-10-20 (Estimated); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Non-small Cell Lung Cancer
Keywords: invasive staging; mediastinal lymph nodes; endosonography; surgical staging; lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thoracic endosonography (Experimental): Endobronchial-ultrasound controlled transbronchial needle aspiration (EBUS-TBNA) in combination with a transoesophageal-ultrasound controlled needle aspiration of mediastinal lymph nodes
  Interventions: Procedure: Thoracic endosonography

INTERVENTIONS:
Procedure: Thoracic endosonography — Endobronchial-ultrasound controlled transbronchial needle aspiration (EBUS-TBNA) in combination with a transoesophageal-ultrasound controlled needle aspiration of mediastinal lymph nodes
  Other Names: thoracic echo-endoscopy

SUMMARY:
This is a prospective non-randomized multicenter clinical trial performing endobronchial and esophageal ultrasound for mediastinal lymph node staging of operable and resectable cT1-T2-selectedT3 cN1 cM0 NSCLC.

DETAILED DESCRIPTION:
Provided no mediastinal lymph node metastases are proven by echoendoscopy, all patients will subsequently undergo surgical staging. Patients without tissue proof of mediastinal nodal disease at surgical staging will undergo a thoracotomy with systematic lymph node dissection. Provided mediastinal lymph node metastases are proven by echoendoscopy, the patient goes off study protocol and can further be assessed/treated according to local clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with operable and resectable (suspected) NSCLC
* Patients with clinical N1 staging based on PET/CT
* Only T1, T2, and selected T3 (i.e. intraparenchymal tumour >7cm, chest wall, or additional nodule in the same lobe) are allowed.

Exclusion Criteria:

* Patients with enlarged mediastinal lymph nodes on chest CT or FDG-PET positive mediastinal lymph nodes
* Patients with a central tumour staged T3 or any T4.
* All stage IV patients.
* Patient unable to give informed consent.
* Patient previously underwent a mediastinoscopy.
* Tracheal or upper airway stenosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-01; Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of echo-endoscopic mediastinal staging in operable and resectable cT1-2-selectedT3 cN1 NSCLC | One month

SECONDARY OUTCOMES:
NPV of echo-endoscopic mediastinal staging in operable and resectable cT1-2-selectedT3 cN1 NSCLC | one month
Cost-effectiveness analysis for echo-endoscopy in cN1 disease NSCLC | one month

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Dooms, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Kurt Tournoy, Principal Investigator — University Ghent
Locations (3):
- Belgium (2):
  - Universitair Ziekenhuis Gent, Ghent
  - Universitaire Ziekenhuizen leuven, Leuven
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Derived] Dooms C, Tournoy KG, Schuurbiers O, Decaluwe H, De Ryck F, Verhagen A, Beelen R, van der Heijden E, De Leyn P. Endosonography for mediastinal nodal staging of clinical N1 non-small cell lung cancer: a prospective multicenter study. Chest. 2015 Jan;147(1):209-215. doi: 10.1378/chest.14-0534. PMID 25211526